CLINICAL TRIAL: NCT03178578
Title: A Prospective Observational Study of the Expectations and Physiological Effects of Fluid Bolus Therapy in the Intensive Care Unit
Brief Title: A Prospective Observational Study of the Expectations and Physiological Effects of Fluid Bolus Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Austin Hospital, Melbourne Australia (Other); Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Christer Svensen, Professor, Karolinska Institutet
Other Study IDs: LNR/17/Austin/94
Record Dates: First submitted 2017-04-21; First posted 2017-06-07 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Hypovolemia; Sepsis; Post-operative Hypovolemia; Fluid Therapy
Keywords: Fluid therapy
MeSH Terms: conditions — Hypovolemia; Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study aims to (i) asses intensive care doctors trigger for and the expected physiological response to a fluid bolus and (ii) evaluate the patient's actual physiological response to a single fluid bolus at one hour post-bolus for 100 adult patients admitted to the intensive care unit will be included in the study.

DETAILED DESCRIPTION:
Intensive care unit patients often receive a fluid bolus during their ICU-stay. ICU doctors use a variety of clinical triggers when deciding whether or not to give a fluid bolus. However, the type of physiological triggers used and their correlation to the anticipated physiological response of the patient to an administered fluid bolus is not entirely clear.

The investigators will perform a prospective observational study to evaluate the triggers for, expected physiological and actual physiological response to fluid bolus therapy in the intensive care unit. Specifically, the investigators will assess which of the the physiological trigger(s) intensive care doctors use when deciding to give a fluid bolus; the expected physiological response to the fluid bolus by intensive care doctors; and, to what degree the patients actual physiological response 1 hour after a fluid bolus correlate with expectations.

This study will involve a survey of ICU physicians to determine the physiological trigger and expectations and a medical audit to ascertain the physiological response to a fluid bolus. The investigators will evaluate a single fluid bolus in 100 separate intensive care unit patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the intensive care unit and prescribed a fluid bolus.

Exclusion Criteria:

* The intensive care physician declines to participate.
* Expected survival < 24h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypovolemic critically ill patients in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-18 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of anticipated hemodynamic effects at completion of bolus | At completion of bolus
  The accuracy and precision between the expected and the observed physiological effects will be described using Bland-Altman methodology

SECONDARY OUTCOMES:
Accuracy of anticipated hemodynamic effects at one hour after completion of the fluid bolus | At one hour after completion of the fluid bolus
  The accuracy and precision between the expected and the observed physiological effects will be described using Bland-Altman methodology
The hemodynamic effects of a fluid bolus at completion of bolus | At completion of bolus
  The effect of the fluid bolus on blood pressure at completion of bolus will be described.
The hemodynamic effects of a fluid bolus at one hour after completion of the fluid bolus | At one hour after completion of the fluid bolus
  The effect of the fluid bolus on blood pressure one hour after completion of the fluid bolus will be described.
The hemodynamic effects of a fluid bolus at completion of bolus | At completion of bolus
  The effect of the fluid bolus on heart rate at completion of bolus will be described.
The hemodynamic effects of a fluid bolus at one hour after completion of the fluid bolus | At one hour after completion of the fluid bolus
  The effect of the fluid bolus on heart rate one hour after completion of the fluid bolus will be described.
The hemodynamic effects of a fluid bolus at completion of bolus | At completion of bolus
  The effect of the fluid bolus on cardiac index at completion of bolus will be described.
The hemodynamic effects of a fluid bolus at one hour after completion of the fluid bolus | At one hour after completion of the fluid bolus
  The effect of the fluid bolus on cardiac index one hour after completion of the fluid bolus will be described.
The hemodynamic effects of a fluid bolus at completion of bolus | At completion of bolus
  The effect of the fluid bolus on CVP at completion of bolus will be described.
The hemodynamic effects of a fluid bolus at one hour after completion of the fluid bolus | At one hour after completion of the fluid bolus
  The effect of the fluid bolus on CVP one hour after completion of the fluid bolus will be described.
The hemodynamic effects of a fluid bolus at completion of bolus | At completion of bolus
  The effect of the fluid bolus on ScVO2 or SvO2 at completion of bolus will be described.
The hemodynamic effects of a fluid bolus at one hour after completion of the fluid bolus | At one hour after completion of the fluid bolus
  The effect of the fluid bolus on ScVO2 or SvO2 one hour after completion of the fluid bolus will be described.
The hemodynamic effects of a fluid bolus at completion of bolus | At completion of bolus
  The effect of the fluid bolus on lactate levels at completion of bolus will be described.
The hemodynamic effects of a fluid bolus at one hour after completion of the fluid bolus | At one hour after completion of the fluid bolus
  The effect of the fluid bolus on lactate levels one hour after completion of the fluid bolus will be described.
The hemodynamic effects of a fluid bolus at completion of bolus | At completion of bolus
  The effect of the fluid bolus on urine output at completion of bolus will be described.
The hemodynamic effects of a fluid bolus at one hour after completion of the fluid bolus | At one hour after completion of the fluid bolus
  The effect of the fluid bolus on urine output one hour after completion of the fluid bolus will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Christer Svensen, MD,PhD,Prof, Principal Investigator — Karolinska Institutet
Locations (3):
- Austin Hospital, Melbourne, Victoria, Australia
- Sweden (2):
  - Danderyds sjukhus, Stockholm, Danderyd
  - Södersjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: No